CLINICAL TRIAL: NCT01281280
Title: A Post-Market, Open Observational Long-term Effectiveness Follow-up Study of Participants With Drug-resistant Epilepsy With Partial-onset Seizures Previously Enrolled in a Randomized Controlled Trial (E-100: PuLsE) Comparing Best Medical Practice With or w/o Adjunctive Vagus Nerve Stimulation Therapy
Brief Title: PuLsE 2-Observational Long-Term Effectiveness Follow-Up Study of PuLsE 1
Acronym: PuLsE 2
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Epilepsy (E)-101; E-101 PuLsE 2 (Other: Cyberonics)
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Epilepsy
Keywords: PuLsE 2, Drug-resistant Epilepsy Partial-onset Seizures
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VNS Therapy
- Best Medical Practice

SUMMARY:
This is a post-market, open observational long-term effectiveness follow-up study of participants with drug-resistant epilepsy with partial-onset seizures previously enrolled in a randomized controlled trial (PuLsE) comparing Best Medical Practice with or without adjunctive Vagus Nerve Stimulation Therapy.

DETAILED DESCRIPTION:
In 2005 Cyberonics, Inc. initiated PuLsE: an open, prospective, randomized, parallel group study directly comparing Best Medical Practice with and without adjunctive VNS Therapy.

In July 2008, the decision was made to discontinue this study due to lower than expected enrolment, impairing the possibility to meet the primary objective with appropriate statistical power. However, the relatively large number of participants (n=121) randomized in the original PuLsE study offers the possibility to generate scientifically valuable and original findings if additional follow-up data can be gathered. After consultation with the PuLsE Investigators, Cyberonics decided to implement an observational long-term follow-up of the participants enrolled in the original PuLsE study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, the participant must meet all the following criteria:

1. Participant must have been randomized in the original PuLsE study.
2. Participant must have baseline data from the original PuLsE study.
3. Participant is able to give accurate seizure counts, health outcomes information, and complete study instruments with minimal assistance.
4. Participant or legal guardian understands study procedures and has voluntarily signed an informed consent for PuLsE 2 in accordance with institutional and local regulatory policies.

Exclusion Criteria:

The presence of any of the following will exclude a participant from the study:

1. Participant has a history of non-compliance with the completion of a seizure diary.
2. Participant currently uses, or is expected to use during the study, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy.
3. Participant is expected to require full body magnetic resonance imaging during the clinical study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of participants previously enrolled in the original PuLsE study diagnosed with drug-resistant epilepsy with partial-onset seizures. All patients will be analyzed according to the treatment that they have actually received and followed in this new study regardless of what treatment groups they were randomized in the previous study.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Exploratory evaluations | 5 years
  The objective of this post-market study is to perform exploratory evaluations to identify clinically and statistically significant predictors of response at all follow-up visits in participants with drug-resistant epilepsy with partial-onset seizures treated with Best Medical Practice with or without adjunctive VNS Therapy. This will be accomplished through regression modeling of the response variates (including change in baseline quality of life score and percent reduction in seizure frequency).

SECONDARY OUTCOMES:
Change from baseline at all follow-up visits of Best Medical Practice with adjunctive VNS Therapy compared to Best Medical Practice | 5 years
Change from baseline at all follow-up visits across all health outcome measurements | 5 years
Evaluation of safety and tolerability | 5 Years
Evaluation of change from baseline at all follow-up visits of Best Medical Practice with and without adjunctive VNS Therapy on health outcome measurements and quality of life (QOL) | 5 Years
Sub-analysis to evaluate the change from baseline on quality of life | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ryvlin, MD, Principal Investigator — Unité d'épileptologie
Locations (18):
- Belgium (2):
  - ULB Hopital Erasme, Brussels
  - UZ Gent, Ghent
- Canada (2):
  - QE2 Health Sciences Centre Department of Neurology, Halifax
  - Hopital Notre Dame, Montreal
- France (4):
  - CHU Grenoble, Grenoble
  - Hopital Roger Salengro Service de Neurologie, Lille
  - Hopital Neurologique Unite d' epileptologie, Lyon
  - Hopital Gui De Chauliac, Montpellier
- Germany (2):
  - Universitatskliniken Bonn, Bonn
  - Universitatsklinl Erlangen Zentrum fur Epilepsie, Erlangen
- Italy (6):
  - Azienda Ospedaliero Universitaria, Ancona
  - Universita di Bologna, Bologna
  - Universita di Pisa, Pisa
  - Azienda Ospedialiera "Bianchi Melacrino Morelli", Reggio Calabria
  - Unisersita Cattolica Del Sacro Cuore, Rome
  - Centro Epilessia, Torino
- Hans Berger kliniek Neurology, Oosterhout, Netherlands
- The National Hospital for Neurology and Neurosurgery, London, United Kingdom